CLINICAL TRIAL: NCT03672903
Title: Effect of Different Weight Vests on Body Weight in Obese Individuals
Acronym: EVO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EVO
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Obesity
Keywords: obesity; weight vest; gravitostat; appetite; obesity treatment; leptin; body weight; weight loss; diet-induced obesity; osteocytes; glucose metabolism
MeSH Terms: conditions — Obesity; Body Weight; Weight Loss

STUDY DESIGN:
Intervention Model Description: We will use a parallel study design in which we compare the placebo group with the intervention group. In order to avoid the risk of carry-over effects, we have decided to not use a crossover design. This could have decreased the variation of the measurement values and increased the power of the study. However, we believe there could be a risk of a carry-over effect with a cross over design. As this is a completely new effect in clinical studies, we have no information about the wash-out time needed to avoid this problem.
Who Masked: Participant
Masking Description: Masking will not be publically revealed before the study ends. Subjects may be able to determine if they are in the control/placebo group or intervention group if we publically reveal our masking procedure. However, the masking procedure is pre-determined and approved by the ethic's committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects in this arm will carry heavy weight vests for three weeks.
  Interventions: Device: Weight Vest
- Control (Placebo Comparator): Subjects in this arm will carry light weight vests for three weeks.
  Interventions: Device: Weight Vest

INTERVENTIONS:
Device: Weight Vest — A vest with added weights up to a maximum of 15 kg.
  Other Names: artificial weights

SUMMARY:
Obesity related ailments, such as cardiovascular diseases (CVD) and metabolic disorders are major causes of death in the Western World. The proposed research may result in improved prevention, diagnosis and treatments of obesity and obesity-related disorders. Recently published data show that if a weight is carried by a rodent, this animal will lose body weight and gain an improved glucose control.

We aim to confirm these findings in a human model. We plan to let obese subjects carry weight vests and monitor their change in body weight. We will also measure appetite, physical activity and insulin sensitivity to further examine the potential beneficial effects of loading. Blood sampling will be performed to investigate the mechanism of action.

DETAILED DESCRIPTION:
STUDY OBJECTIVES AND ENDPOINTS

Primary objective

To determine if wearing a weight vest with 11 % of an individual's body weight for 3 weeks decreases body weight in obese study subjects.

Secondary objective

To determine if wearing a weight vest with 11 % of an individual's body weight for 3 weeks affects fat mass, bone mass, muscle mass, water mass, fat free mass, physical activity and food intake in obese study subjects.

To determine if wearing a weight vest with 11 % of an individual's body weight for 3 weeks affects plasma concentrations of glucose, insulin, HDL, LDL, TAG, FGF21, osteocalcin, FGF23, FGF15, sclerostin, lipocalin-2, leptin, ghrelin, GLP-1, GLP-2, CCK, (3-36)PYY, glucagon, renin, methoxynorepinephrine, Na, K, Cl, Ca and creatinine.

STUDY DESIGN AND PROCEDURES

Overall study design and procedure protocol

The aim of the study is to investigate the effect of adding synthetic weights to obese individuals. The weights will be added as a weight vest with 11 % of the individual's body weight and will be worn for three weeks. Half of the study subjects will be given a weight vest with 11 % of body weight and half of the study subjects will be given a light weight vest. The light weight vest consists of a weight vest with most of the weights removed. The weight of the light vest will be 1 % of body weight giving a difference of 10 % between the groups.

Body weight, fat mass, bone mass, water mass and fat free mass will be measured before and after the intervention by medical personnel to determine the effect of added synthetic weights on obese subject. This will be measured using bioelectrical impedance analysis (BIA) (MC-180MA, Tanita). The scales will be calibrated every week during the study to make certain reliable measurements.

Pedometers will be used to measure the subject's activity each study day. We will also encourage the study participants to report food intake, choice of food and level of hunger each week. This will be done using the validated poll MiniMealQ(9). A pedometer will also be attached to the vests to check the daily use of the vests. The study persons will be informed about this arrangement.

Fasting blood sampling will be performed before and after the intervention to further determine the effects of adding synthetic weights to obese individuals but also to elucidate the mechanism behind the "gravitostat". Blood glucose levels will be measured immediately. Blood samples, except blood glucose, will be analyzed either continuous or after all study subjects have been enrolled depending on human resources.

Study subjects will be recruited by advertising in the local newspaper. Study subjects will be informed about hypothesis that people carrying a heavy or light weight may differ in weight loss. At this point it is not known if the heavy weight vest or the light vest is causing more weight loss, as no one has performed similar studies on humans.

Study subjects will have one week to familiarize themselves with the equipment used in the study before the intervention starts. This is to minimize human errors during the intervention and ensure a high level of compliance. The data collected during this week will be used as baseline.

Day 1 - enrollment

The first 100 persons to contact the researchers will be enrolled in the study. In order to be enrolled a study subject also need to meet all the inclusion criteria and not meet any of the exclusion criteria. The study subjects will be entitled to a private meeting with one of the researchers. Study subjects will receive information about the study plan both orally and written during this meeting.

Consumption of more than one liter of wine (11 %) or alcohol equivalent during a study week will not be accepted. Drastic change in lifestyle before or during the study will not be accepted. Any study subject failing to comply with this restriction will instantly be removed from the study.

Education and detailed planning of the study subjects will be performed after written consent is obtained from the study subject. Body weight, fat mass, bone mass, water mass and fat free mass will be measured using BIA. It is unlikely that bone mass and water mass will be affected during the short time of this study but these values are easily obtained during the measurements. We will also measure blood pressure, height in order to calculate BMI and collect each subject's age and gender.

This meeting will end with a blood sample to screen for common diseases that may distort the results and increase the risk of adverse effects. We will measure the following substances in blood: hemoglobin, white blood cells, trombocytes, sodium, potassium, creatinine, ASAT, ALAT, HbA1c, C-reactive protein (CRP), T4, TSH. Also, we will use urine dipsticks to further screen for diseases. We will measure the following substances in urine: nitrite, white blood cells, red blood cells, glucose, creatinine and albumin. Only subjects were all above substances are within normal levels will be included in the study.

Study subject will be able to contact the researchers by e-mail or mobile phone any time during the study if questions arise.

Day 8 - intervention starts

Study subjects will be entitled to another appointment with the researchers and the nurse from Gothia Forum one week after the enrollment. Body weight, fat mass, bone mass, fat free mass and water mass will be measured during this meeting using BIA.

Fasting blood sampling by an experienced nurse from Gothia Forum will be performed when the researcher believe that the study subject is fully educated and ready to be enrolled in the study. A maximum of 25 ml will be collected at each blood sampling. Plasma levels of glucose will be measured instantly in capillary blood, and thus not be dependent on successful venous blood sampling. Venous blood samples for other measurement than glucose will be centrifuged by the researchers or personnel from Gothia Forum to obtain serum or EDTA plasma samples. Serum and plasma samples may be stored at a temperature of -80°C until analysis. Study subjects can request to have their blood samples destroyed at any time.

The intervention will start directly after blood sampling. Subjects will earn a randomized three character code to be used throughout the study; this will be noted in a digital only randomization list. Study subjects will obtain either a weight vest with 11 % of body weight or a light vest weighing 1 % of body weight. The vest is to be worn 8 hours each day for the following 3 weeks. The vest is only to be used during awake hours.

Day 15

Study subjects will be entitled to another appointment with the researchers two weeks after the enrollment, this appointment may be performed by telephone if the subject so agree. Any problems with compliance will be discussed. Study subjects who deviate more than 20 % from the study protocol will be removed from the study. Study subjects will continue to wear the vests for 8 hours each day.

Day 22

Study subjects will be entitled to another appointment with the researchers three weeks after the enrollment, this appointment may be performed by telephone if the subject so agree. Any problems with compliance will be discussed. Study subjects who deviate more than 20 % from the study protocol will be removed from the study. Study subjects will continue to wear the vests for 8 hours each day.

Day 29 - intervention ends

Study subjects will be entitled to another appointment in the morning before breakfast with the researchers and the nurse from Gothia Forum four weeks after the enrollment. Body weight, fat mass, bone mass, fat free mass and water mass will be measured during this meeting using BIA. Fasting glucose will be measured in capillary blood. Venous blood sampling will be done. Study subjects will have worn the vests for 8 hours the day before, but they will not wear it during the visit the morning of day 29.

The appointment at day 29 may also be performed on "day 30" depending on the study subject's schedule. Nevertheless, last day for the intervention is on study day 29.

Rationale for study design

In order to avoid the risk of carry-over effects, we have decided to not use a crossover design. This could have decreased the variation of the measurement values and increased the power of the study. However, we believe there could be a risk of a carry-over effect with a cross over design. As this is a completely new effect in clinical studies, we have no information about the wash-out time needed to avoid this problem.

ELIGIBILITY:
Inclusion Criteria:

1. Obesity as defined by a BMI >30 and ≤35. Fat mass should be above 25 %.
2. 18-70 years of age. We will primarily recruit men. Women will only be recruited if we are unable to find 80 eligible male participants.
3. Consent out of free will.
4. Willingness to comply with the study protocol and restrictions of not consuming excessive amounts of alcohol (maximum 1 litre, 11 % or alcohol equivalent for a full week) or using any drugs. Smoking and snuff use is allowed.
5. Normal screening blood- and urine samples. In blood: hemoglobin, white blood cells, trombocytes, sodium, potassium, creatinine, ASAT, ALAT, HbA1c, CRP, T4, TSH. In urine: nitrite, white blood cells, red blood cells, glucose, creatinine and albumin.
6. Signed informed consent.

Exclusion Criteria:

1. Chronic disease that hardens the participation in the study as judged by the investigator.
2. Chronic pain such as pain that is constant and impairs quality of life; for example: severe back, hip and knee pain.
3. Regular consumption of medicine or natural supplements that affect weight, inhibit physical activity or increase the risk of adverse effects as judged by the investigator. The following drugs will not be accepted: β-antagonists, GLP-1-agonists, SGLT2-inhibitors, sulfonylureas, insulin, orlistat, mysimba and bisphosphonates.
4. Gastric by-pass surgery or equivalent.
5. Reduced mobility.
6. Pregnancy: Females of childbearing potential must confirm to use reliable contraception and not suspect to be pregnant. Subjects may be asked to perform a pregnancy test.
7. Change in body weight of 5 kg or greater during the past 3 months or recently started a strict diet. Also, a greater change in body weight than 1.5 kg difference between day 1 and day 8 will not be accepted.
8. Drastic change in lifestyle during the last 3 months; for example a significant change in physical activity or nicotine, alcohol or drug use.
9. Apparent risk of not being able to comply with the study protocol for any reason as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Body Weight | 3 weeks
  Change in body weight between start of the intervention and end of the intervention, indirectly measuring change in BMI

SECONDARY OUTCOMES:
Appetite | 3 weeks
  Calories consumed and choice of food
Physical Activity | 3 weeks
  Steps taken and walking distance
Metabolism | 3 weeks
  We will measure the change in serum concentration of Na
Metabolism | 3 weeks
  We will measure the change in serum concentration of K
Metabolism | 3 weeks
  We will measure the change in serum concentration of Cl
Metabolism | 3 weeks
  We will measure the change in serum concentration of Ca
Metabolism | 3 weeks
  We will measure the change in serum concentration of Creatinine
Metabolism | 3 weeks
  We will measure the change in serum concentration of insulin
Metabolism | 3 weeks
  We will measure the change in serum concentration of HDL-Cholesterol
Metabolism | 3 weeks
  We will measure the change in serum concentration of LDL-Cholesterol
Metabolism | 3 weeks
  We will measure the change in serum concentration of triacylglycerol (TAG)
Metabolism | 3 weeks
  We will measure the change in serum concentration of FGF21
Metabolism | 3 weeks
  We will measure the change in serum concentration of osteocalcin
Metabolism | 3 weeks
  We will measure the change in serum concentration of FGF23
Metabolism | 3 weeks
  We will measure the change in serum concentration of FGF15
Metabolism | 3 weeks
  We will measure the change in serum concentration of sclerostin
Metabolism | 3 weeks
  We will measure the change in serum concentration of lipocaline
Metabolism | 3 weeks
  We will measure the change in serum concentration of leptin
Metabolism | 3 weeks
  We will measure the change in serum concentration of ghrelin
Metabolism | 3 weeks
  We will measure the change in serum concentration of GLP-1
Metabolism | 3 weeks
  We will measure the change in serum concentration of GLP-2
Metabolism | 3 weeks
  We will measure the change in serum concentration of CCK
Metabolism | 3 weeks
  We will measure the change in serum concentration of (3-36)PYY
Metabolism | 3 weeks
  We will measure the change in serum concentration of glucagon
Metabolism | 3 weeks
  We will measure the change in serum concentration of testosterone
Metabolism | 3 weeks
  We will measure the change in serum concentration of estrogens
Metabolism | 3 weeks
  We will measure the change in serum concentration of renin
Metabolism | 3 weeks
  We will measure the change in serum concentration of methoxynorepinephrine
Fat Mass | 3 weeks
  Change in fat mass between start of the intervention and end of the intervention
Muscle Mass | 3 weeks
  Change in muscle mass between start of the intervention and end of the intervention
Water Mass | 3 weeks
  Change in water mass between start of the intervention and end of the intervention
Bone Mass | 3 weeks
  Change in bone mass between start of the intervention and end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ander Jansson, MD, PhD, Professor, Principal Investigator — Clinical Trial Center, Sahlgrenska University hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jansson JO, Palsdottir V, Hagg DA, Schele E, Dickson SL, Anesten F, Bake T, Montelius M, Bellman J, Johansson ME, Cone RD, Drucker DJ, Wu J, Aleksic B, Tornqvist AE, Sjogren K, Gustafsson JA, Windahl SH, Ohlsson C. Body weight homeostat that regulates fat mass independently of leptin in rats and mice. Proc Natl Acad Sci U S A. 2018 Jan 9;115(2):427-432. doi: 10.1073/pnas.1715687114. Epub 2017 Dec 26. PMID 29279372